CLINICAL TRIAL: NCT04562584
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Brief Title: Pulse Oximeter Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MyHomeDoc Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VVD-MHD-155
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Oximetry
Keywords: myhomedoc; pulse oximetry; oximeter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MyHomeDoc (Experimental): Comparison of MyHomeDoc pulse oximetry readings with arterial blood saturation laboratory analysis in the same subject
  Interventions: Device: MyHomeDoc

INTERVENTIONS:
Device: MyHomeDoc — MyHomeDoc device SpO2 measurements and parallel blood gas analysis to determine oxyhemoglobin saturation (SaO2) using an ABL-90 multi-wavelength oximeter.

SUMMARY:
The aim of this project is to test the accuracy of pulse oximeters (devices intended to measure oxygen saturation in blood noninvasively) during mild, moderate and severe hypoxia (a lower-than-normal concentration of oxygen in arterial blood); ie, a range of arterial HbO2 saturations from 100 to down to 70%. This is done by comparing the reading of the pulse oximeter during brief, steady state hypoxia with a gold-standard measurement of blood oxyhemoglobin (hemoglobin carrying oxygen) saturation, that is arterial blood sample processed in a laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, aged ≥18 and <50.
2. The subject is in good general health with no evidence of any medical problems.
3. The subject is fluent in both written and spoken English.
4. The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. The subject is obese (BMI>30).
2. The subject has a known history of heart disease, lung disease, kidney or liver disease.
3. Diagnosis of asthma, sleep apnea, or use of CPAP.
4. Subject has diabetes.
5. Subject has a clotting disorder.
6. The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
7. The subject has any other serious systemic illness.
8. The subject is a current smoker.
9. Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
10. The subject has a history of fainting or vasovagal response.
11. The subject has a history of sensitivity to local anesthesia.
12. The subject has a diagnosis of Raynaud's disease.
13. The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
14. The subject is pregnant, lactating or trying to get pregnant.
15. The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
16. The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Saturation level measurement | 1 hour
  Induction of hypoxia by having subjects breathe mixtures of nitrogen, room air, and carbon dioxide to allow measurement of oxyhemoglobin saturation between 70-100%. Each plateau level of oxyhemoglobin saturation was maintained for at least 30 seconds or until reference pulse oximeters readings were stable

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Bickler, Ph.D., M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Hypoxia Research Laboratory Department of Anesthesia and Perioperative Care University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No